CLINICAL TRIAL: NCT02688504
Title: CESIR-U2 : Influence of Drugs Use and Health Status
Brief Title: Health and Road Safety: Influence of Drugs Use and Health Status
Acronym: CESIR-U2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/33
Record Dates: First submitted 2015-12-30; First posted 2016-02-23 (Estimated); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Car Accident
Keywords: labelled medicines; drivers involved in serious and non-serious road accidents; relevance and effectiveness of pictograms on medicines packaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- serious road accidents: Drivers involved in serious road accidents (hospitalization > 24 hours)
- non-serious road accidents: drivers involved in non-serious road accidents (hospitalization < 24 hours).

SUMMARY:
In France, drugs affecting driving ability directly or by indicating at-risk diseases are classified in a 4-level standardized classification associated with a graded pictogram.

When the French authorities required this graded pictogram, they commissioned the CESIR-U1 study, a study designed to describe the use of labelled medicines by drivers involved in serious road accidents (hospitalization > 24h). This study, conducted in Bordeaux, Limoges and Toulouse, recruited 679 drivers involved in serious road accidents. When the responsibility of the driver is taken into account, it appears that the association of risk factors (alcohol, sleep, ...) and the use of labelled drugs increases this responsibility. Even though labelled medicines seemed slightly more at risk than unlabelled ones, this did not reach significance.

This conclusion is different from the conclusion of CESIR-A, a data linkage study of the police and the health insurance databases which showed a correlation between the use of grade 2 or 3 labelled medicines and driver responsibility.

This difference between CESIR-U and CESIR-A could be related to a lack of power or to the characteristics of the subjects included (mostly young men and motorcycle drivers). That is why it was thought interesting to increase the size of the sample and to include non serious road accidents (hospitalization < 24 hours) that represent around 73% of accidents.

ELIGIBILITY:
Inclusion Criteria:

* Driver involved in a road accident and admitted in an emergency department
* Aged over 18 years
* Able to respond to a structured questionnaire
* Having agreed to participate in the study

Exclusion Criteria:

* Minors
* Passenger
* Pedestrian
* Discharge or transfer to another hospital/clinic before the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multicentre observational study that will include 2 populations: drivers involved in serious road accidents (hospitalization > 24 hours) and non-serious road accidents (hospitalization < 24 hours). The drivers involved in road accidents and admitted in an emergency department will be identified during daily visits (except on week end) by Clinical Research Associates (CRA) of the different centres. As soon as possible, a structured validated interview will done by a trained CRA.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Drugs use reported by drivers involved in road accidents | inclusion date
  Drugs use is collected during a structured interview administered by a trained CRA. Measure title : percentage of drivers who take drugs, by ATC classification, by pictogram and by drug.

SECONDARY OUTCOMES:
Responsibility of the driver for the accident | inclusion date
  The responsibility of the driver (responsible or not responsible) is a data extracted from the BAAC sheet (a sheet fulfilled by the police in case of traffic crashes)
Seriousness of the accident | inclusion date
  The seriousness of the accident is assessed according the duration of hospital stay. If the duration is less than 24 hours, accidents are considered as non serious. If not, accidents are considered as serious.
Knowledge of drivers about graded pictogram featured on drugs packaging | inclusion date
  Knowledge about graded pictogram is collected during a structured interview administered by a trained CRA. Measure title : percentage of drivers who know if a pictogram is featured on their drugs packagings.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas MOORE, Pr, Study Chair — Plateforme BPE
Locations (2):
- France (2):
  - Hôpital Pellegrin, Bordeaux
  - CH de Perigueux, Périgueux